CLINICAL TRIAL: NCT05353712
Title: Effect of Consuming Products Containing Rare Sugars Alongside Sucrose on Glycaemic Response in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22013
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Glycaemic Response in Healthy Participants
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group T: ABCDEF (Experimental): Participants will receive all six blind-coded samples, in the order A, B, C, D, E, F. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40
- Group V: FABCDE (Experimental): Participants will receive all six blind-coded samples, in the order F, A, B, C, D, E. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40
- Group W: EFABCD (Experimental): Participants will receive all six blind-coded samples, in the order E, F, A, B, C, D. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40
- Group X: DEFABC (Experimental): Participants will receive all six blind-coded samples, in the order D, E, F, A, B, C. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40
- Group Y: CDEFAB (Experimental): Participants will receive all six blind-coded samples, in the order C, D, E, F, A, B. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40
- Group Z: BCDEFA (Experimental): Participants will receive all six blind-coded samples, in the order B, C, D, E, F, A. There will be a minimum of 7 days washout between samples.
  Interventions: Other: SUCROSE; Other: CONTROL; Other: ARA20; Other: ARA40; Other: TAG20; Other: TAG40

INTERVENTIONS:
Other: SUCROSE — 50g sweet creme composed of 14.3g vegetable fat and 35.7g sucrose.
Other: CONTROL — 35.7g sweet creme composed of 14.3g vegetable fat and 21.4g sucrose.
Other: ARA20 — 42.9g sweet creme composed of 14.3g vegetable fat, 21.4g sucrose and 7.1g L-arabinose
Other: ARA40 — 50g sweet creme composed of 14.3g vegetable fat, 21.4g sucrose and 14.3g L-arabinose
Other: TAG20 — 42.9g sweet creme composed of 14.3g vegetable fat, 21.4g sucrose and 7.1g D-tagatose
Other: TAG40 — 50g sweet creme composed of 14.3g vegetable fat, 21.4g sucrose and 14.3g L-arabinose

SUMMARY:
Food manufacturers are being tasked to reduce the added sugar content of products. Rare, but natural sugars, may serve as useful sweeteners as they are low-calorie, safe, sweet and have a mild taste. Previous studies have shown that consuming rare sugars alongside other carbohydrates leads to a lower spike in blood glucose after eating. This means that products containing rare sugars may provide health benefits. However, most studies use rare sugars in a glucose drink, so the effect of consuming rare sugars in foods is not known.

The aim of this study is to find out whether consuming sweet crème products containing rare sugars reduces the blood glucose response compared to sucrose-only products. The effect of the rare sugar products on hunger and appetite will also be assessed.

Participants will attend the Clinical Research Facility on 6 occasions, after fasting for 10 hours. At each visit, they will consume a different sample of sweet crème. They will be asked to give blood samples before eating the sample, and at regular intervals for 2 hours afterwards. They will also complete questionnaires to assess their appetite using linear scales. Blood samples will be analysed in the laboratory to measure the level of glucose and insulin at each time point. The changes in blood glucose and insulin after consuming the different samples will be compared to find out if the samples containing rare sugars reduced the response.

DETAILED DESCRIPTION:
Main Hypotheses:

This study is designed to test two main hypotheses:

1. Sweet crème products containing the rare sugars arabinose or tagatose will cause a lower spike in blood glucose and insulin than sucrose-only products.
2. Sweet crème products containing the rare sugars arabinose or tagatose will be no less satiating than sucrose-only products.

The null hypotheses are therefore:

1. Levels of blood glucose and insulin are not significantly different after consuming sweet crème products containing rare sugars compared to sucrose-only products.
2. Appetite and food intake are significantly higher after consuming sweet crème products containing rare sugars compared to sucrose-only products.

Study Overview:

This study will be a double-blind crossover trial, allowing each participant to act as their own control. Twenty participants will be recruited and fully informed about the study before giving informed consent. Eligible participants will attend the Clinical Research Facility on 6 separate mornings following an overnight fast. On each occasion participants will consume 40-50g of sweet crème served with commercially available sweet wafers. Sweet crème samples will contain vegetable fat and sucrose with or without the addition of D-tagatose or L-arabinose. Neither the participants or the researchers administering the tests will be aware of which sample is being consumed at each visit. Blood samples will be taken before consumption and at regular intervals for 120 minutes afterwards. Blood samples will be analysed to measure plasma glucose, insulin, and the appetite-regulating hormones GLP-1 and GIP. During each visit participants will also be asked to complete questionnaires assessing their hunger and desire to eat, and any gastrointestinal symptoms.

Samples:

Six different sweet crème samples will be included as listed below:

SUC- Full-sucrose sample (2.5:1 sucrose:vegetable fat)

CONTROL- Reduced-sucrose sample (1.5:1 sucrose:fat)

ARA20- Low-dose arabinose sample (1.5:1:0.5 sucrose:fat:arabinose)

ARA40- High-dose arabinose sample (1.5:1:1 sucrose:fat:arabinose)

TAG20- Low-dose tagatose sample (1.5:1:0.5 sucrose:fat:tagatose)

TAG40- High-dose tagatose sample (1.5:1:1 sucrose:fat:tagatose)

Using these samples, we will be able to investigate the effect of adding rare sugars to a constant sucrose/fat load (by comparing each experimental product with the control product), and also to investigate the effect of replacing sucrose with rare sugars (by comparing ARA40 and TAG40 products with the SUC product).

Study visits:

Each participant will visit on 6 occasions and consume one of the six samples on each visit in a randomised order.

Visits will be separated by at least one week, so each participant is expected to be involved in the study for 2-3 months from start to finish. A randomised crossover design has been selected so that each participant can act as their own control, which reduces the impact of variation in glycaemic response between individuals. The crossover design will therefore allow us to detect significant differences with a smaller number of participants.

At each clinic visit we will measure the glycaemic response (increase in blood glucose and insulin), using methods similar to the standard methodology for assessing glycaemic index. We will also evaluate the effect of the samples on hunger and desire to eat, and gastrointestinal symptoms, using adapted validated questionnaires.

The procedures for each clinic visit are summarised below:

1. Pre-visit fast:

   Participants will fast for 10 hours before visit. All visits will be scheduled before 10am.
2. Clinic visits:

   Participants will visit the clinic on 6 occasions, separated by at least one week. Each visit will last around 3 hours. Every effort will be made to ensure participants are comfortable during clinic visits. Participants will be seated comfortably throughout, and will be asked to remain seated as much as possible. They will be allowed to read or use laptops/phones, and toilet visits will be permitted.
3. Health questionnaire:

   An initial health questionnaire will ask for details of BMI, smoking, alcohol consumption, habitual exercise and gastrointestinal symptoms. Questionnaires on subsequent visits will assess gastrointestinal symptoms only.
4. Blood sampling:

   Research nurses at the CRF will insert cannula in a vein in the hand. Blood will be sampled at baseline and at 15, 30, 45, 60, 90 and 120 minutes after consumption of the sample.
5. Consumption of product and sensory question:

   Researchers will ask participants to consume a sample consisting of 40-50g sweet crème served with commercially available wafers. They will be asked to rate their liking of the product on a 9-point hedonic scale.

   The quantity and composition of the samples has been carefully considered to ensure that they will cause a sufficient glycaemic response for us to be able to detect significant differences between samples. The composition is similar to typical sweet crème products (eg the centre of an Oreo biscuit), and it will be served with ice cream wafers to increase the palatability for participants. Participants will be asked to rate their liking of each sample immediately after consuming it using a hedonic scale.

   Neither the participant nor the researcher administering the clinic visit will be aware of which sample is being consumed at each visit.
6. Appetite questionnaires:

   Researchers will administer paper-based questionnaires using visual analogue scores to ask participants how hungry/full they feel and their desire to eat certain foods. In order to capture changes in appetite over the clinic visit, participants will be asked to complete the same questionnaire at baseline and at 35, 65 and 125 minutes after consuming the product.
7. Buffet meal:

   After the 120 minute blood sampling, cannulas will be removed and participants will be offered a buffet meal consisting of a range of sweet and savoury foods, served with water. Researchers will record the food intake of each participant.
8. 24 hour food diary: Participants will be asked to record their food intake for the rest of the day (until midnight on the day of the study visit) on a paper-based food diary.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of any gender and any sociodemographic background, who are capable of giving informed consent.
* Aged 18 years or over (no upper age limit).
* Able to understand spoken and written English well enough to understand the consent forms and information sheets, and to give responses to questionnaires.

Exclusion Criteria:

* Diagnosed hyperglycaemia, insulin resistance, diabetes or high blood pressure.
* Allergy, intolerance, sensitivity or dietary restriction that would prevent the consumption of the sweet crème samples.
* Anxiety/phobias that would prevent the sampling of venous blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Integrated area under the curve (iAUC) for plasma glucose. | 120 minutes
  Differences in the iAUC for plasma glucose after consuming each product.

SECONDARY OUTCOMES:
Peak plasma glucose | 120 minutes
  Differences in the peak value for plasma glucose after consuming each product.
Integrated area under the curve (iAUC) for plasma insulin. | 120 minutes.
  Differences in the iAUC for plasma insulin after consuming each product.
Peak plasma insulin | 120 minutes.
  Differences in the peak value for plasma insulin after consuming each product.
Integrated area under the curve (iAUC) and peak value for plasma GLP-1. | 120 minutes.
  Differences in the iAUC and peak value for plasma GLP-1 after consuming each product.
Integrated area under the curve (iAUC) and peak value for plasma GIP. | 120 minutes.
  Differences in the iAUC and peak value for plasma GIP after consuming each product.
Food intake at ad libitum buffet meal | 60 minutes
  Total energy intake, macronutrient intake at ad libitum meal 120 minutes after product consumption.
24 hour food intake | 24 hours
  Total energy intake, macronutrient intake until midnight after product consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Jethwa, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - University of Nottingham, Loughborough, Leicestershire
  - Clinical Research Facility, Medical School, University of Nottingham, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No